CLINICAL TRIAL: NCT03837093
Title: A Study of the Dose-response Relationship of Low-dose IL-2 to the Kinetics of Regulatory T-cell Response in Healthy Volunteers
Brief Title: Low-dose IL-2 to the Kinetics of Regulatory T-cell in Healthy Volunteers
Acronym: HEALTHIL-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: APHP180274; 2018-004123-37 (EudraCT Number); MEDAECNAT-2018-11-0048 (Other: ANSM); 2-17-33 (Other: CPP)
Record Dates: First submitted 2019-01-17; First posted 2019-02-11 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
Keywords: Low dose of IL-2; Healthy volunteers; Kinetic study
MeSH Terms: interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- dose A (Experimental): ILT-101
  Interventions: Drug: ILT101
- dose B (Experimental): ILT-101
  Interventions: Drug: ILT101
- dose C (Experimental): ILT-101
  Interventions: Drug: ILT101
- dose D (Experimental): ILT-101
  Interventions: Drug: ILT101
- dose E (Experimental): ILT-101
  Interventions: Drug: ILT101
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ILT101 — Subcutaneous injections starting with induction course with once-daily administration for 5 consecutive days, followed by maintenance course with once every weeks administration during three weeks
  Other Names: low-dose IL-2
  Arms: dose A; dose B; dose C; dose D; dose E
Drug: Placebo — Subcutaneous injections starting with induction course with once-daily administration for 5 consecutive days, followed by maintenance course with once every weeks administration during three weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and the dose-response relationship of ILT-101 to blood Tregs.

DETAILED DESCRIPTION:
In the healthy physiological state, there is homeostasis between regulatory T cells (Tregs) and effector T cells (Teffs) which is deregulated in autoimmune diseases (AID).

The existence of an AID indicates a lack of Tregs. Our team has discovered that low-dose interleukin-2 (ld-IL2) activates and specifically increases Tregs in humans and thus may improve AID. Exploiting this potential requires i) to better target the dose with the best benefit / risk ratio and also ii) to better understand the mechanism of action of this molecule through clinical trials of ld-IL2 in progress, including in type 1 diabetes, multiple sclerosis and systemic lupus erythematosus. During these clinical trials, a very thorough immunological follow-up is carried out in order to discover biomarkers of treatment efficacy. Exploitation of these results will benefit both the cross-analysis of the effects of IL-2 in these 3 diseases with distinct pathophysiologies, but also very importantly a comparison with the effects of ld-IL2 at the healthy volunteer. These analyzes should make it possible to define the most effective dose of IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Without any chronic diseases diagnosed (including allergies);
* Effective contraception> 2 weeks before the first administration of the experimental drug or its placebo and β-hCG negative at the verification of the selection criteria;
* Affiliated to a social security system;
* Free, informed and written consent, signed by the subject and the investigator, before any action required by the research.
* Not taking any treatment

Exclusion Criteria:

* Subject in a period of exclusion of participation in other biomedical research;
* Participation in another research ≤ 1 month and during the study except for research Transimmunom (Non-interventional research involving the human person);
* known antecedents of autoimmune diseases;
* Hypersensitivity to any of the excipients of the investigational drug (mannitol, sodium laurilsulfate, monosodium phosphate dihydrate, disodium phosphate dihydrate);
* Evolutionary infection requiring treatment;
* Viral infection and benign infection less than 2 months old;
* Venous capital not allowing blood samples;
* Pregnant or lactating women;
* Men and women of childbearing potential without effective contraception during the study;
* Live attenuated virus vaccination in the month prior to inclusion or during the study;
* Surgical intervention ≤ 2 months or planned during the study;
* Psychiatric pathology or drug addiction that may impair ability to comply with protocol requirements or give informed consent;
* Presence or history of cancer that has not been cured for less than 5 years, except in situ cervical cancer, or basocellular cancer;
* Subject under a legal protection measure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Variation of Tregs(in (expressed in % of CD4 and total) | from Day 1 to Day 5

SECONDARY OUTCOMES:
AUC corresponding to the évolution of residual values of tregs/CD4+ | Day 5 to Day 60
numbers of different circulating immune populations | baseline to Day 60
levels of serum cytokine(pg) | from baseline to Day 60
levels of serum chemokine | from baseline to Day 60
composition of the intestinal microbiota | from baseline to Day 60
adverse events, anti IL-2 autoantibodies | from baseline to Day 60
levels of serum anti-IL-2 autoantibodies | from baseline to Day 60

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, MD, Principal Investigator — Investigation Center in Biotherapy et immunology Hôpital Universitaire Pitié-Salpêtrière 83 bd de l'Hôpital 75013 Paris l'hopital 75013 Paris; Roberta Lorenzon, MD, Study Director — Clinical Investigation Center Paris Est Hôpital Universitaire Pitié-Salpêtrière 83 bd de l'Hôpital 75013 Paris
Locations (1):
- Clinical Investigation Center Paris Est Hôpital Universitaire Pitié-Salpêtrière 83 bd de l'Hôpital 75013 Paris, Paris, France